CLINICAL TRIAL: NCT06664554
Title: Predictive Value of Maternal Blood Protein Signatures in Preterm Birth
Status: Completed | Type: Observational
Sponsor: HBI Solutions Inc. (Industry)
Collaborators: Shenzhen Maternity & Child Healthcare Hospital (Other)
Responsible Party: Principal Investigator, Qiong Luo, M.D., Ph.D., Women's Hospital School Of Medicine Zhejiang University
Other Study IDs: PTB_01
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Preterm Birth
Keywords: Preterm birth; Maternal blood; Serological protein
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Preterm birth: Pregnancy with delivery before 37 weeks of gestational age
- Term birth control: Pregnancy with delivery at 37 weeks or later of gestational age

SUMMARY:
Accurate prediction of preterm birth is critical for clinical management to improve the neonatal and maternal outcomes. A clinical challenge remains for current predicting biomarkers due to the complexity and multifactorial nature of underlying causes of preterm birth.

This study aims to evaluate the prediction performance of new maternal blood biomarkers (proteomic markers) on the occurrence of preterm birth.

DETAILED DESCRIPTION:
Preterm birth (PTB), defined by delivery before 37 weeks of gestational age, represents a substantial public health challenge due to its elevated rates of neonatal morbidity and mortality worldwide. The prevalence of PTB exhibits variation, ranging from approximately 12-13% in the USA to 5-9% in other developed nations, underscoring a complex issue marked by regional disparities.

Emphasizing its significant public health ramifications, PTB is recognized as a primary contributor to mortality among children under five, particularly with 40% of deaths occurring within the first month of life in this demographic. Following PTB, infants face an increased vulnerability to severe complications like respiratory distress syndrome, intraventricular hemorrhage, and necrotizing enterocolitis, accentuating the acute threats to infant well-being and longevity. Addressing these early-life hurdles requires the formulation of robust strategies for prediction and prevention to alleviate the immediate hazards linked with premature birth.

Preventing PTB crucially depends on accurately identifying women at high risk. Interventions like vaginal progesterone and cervical cerclage are recommended for those with a short cervical length. However, the effectiveness of these strategies is frequently compromised by limitations in current screening methods, which struggle to accurately predict PTB. This underscores a significant gap in effectively identifying all at-risk women, underscoring the necessity for enhanced screening techniques to more precisely pinpoint women who would benefit from preventive interventions.

Current screening methods, primarily based on measuring cervical length and assessing historical risk factors, are inadequate in capturing the multifaceted nature of PTB risk, leading to missed opportunities for intervention and prevention. This inadequacy underscores the importance of developing methods that can more accurately identify women at high risk. Research efforts aimed at addressing these challenges suggest the potential of integrating new biomarkers and maternal characteristics into screening protocols to improve the predictive accuracy of PTB screenings.

Building upon the premise that the placenta plays a pivotal role in fetal health regulation, and that insights into the pathologic mechanisms leading to spontaneous preterm birth can be gleaned from the placental transcriptome, the investigators utilized existing transcriptomic data from the public domain, employing bioinformatics methodologies. This data was further complemented by quantitative proteomics analysis techniques using mass spectrometry. Through this integrated approach, the investigators have developed a novel PTB screening panel comprising three protein biomarkers. The efficacy and prediction performance of this three-protein predictor will be evaluated in this study with independent cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between18 and 45 years of age
* Single pregnancy
* Consent to participate in the study

Exclusion Criteria:

* Premature rupture of membranes
* Uterine malformation
* Fetal malformation
* Pregestational Diabetes
* Systemic diseases (chronic kidney disease, autoimmune disease, etc.)
* Serious medical illness (renal insufficiency, congestive heart disease, chronic respiratory insufficiency, etc.).
* Suffering from other disease unfavorable to the trial such as metal illness
* Any maternal or fetal condition that requires termination of pregnancy.
* Active vaginal bleeding.
* Multifetal pregnancy with greater than or equal to 2 fetuses.
* Lack of clinical outcome or incomplete basic information
* Iatrogenic premature delivery or induced labor
* Lack of consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: General women with pregnancy
Sampling Method: Probability Sample
Enrollment: 18000 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Prediction of preterm birth | After blood draw during doctor's visit before 37 weeks of gestation
  The primary outcome is the prediction of preterm birth, defined as pregnancy duration of less than 37 weeks. Preterm birth prediction score is calculated as sum of the z-score of 3 proteins' multiple of median (MoM) values.

SECONDARY OUTCOMES:
Sensitivity, Specificity, Positive predictive value (PPV), Negative predictive value (NPV) | After blood draw during doctor's visit before 37 weeks of gestation
  Sensitivity, Specificity, PPV and NPV was calculate for identification the preterm birth cases using pre-defined threshold of prediction score.

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Luo, M.D. Ph.D., Principal Investigator — Department of Obstetrics, Women's Hospital of Zhejiang University, School of Medicine, Hangzhou, 310006, China
Locations (5):
- China (5):
  - Department of Obstetrics and Gynecology, the Eighth Affiliated Hospital, Sun Yat-sen University;, Shenzhen, Guangdong
  - Department of Obstetrics, Shenzhen Maternity and Child Healthcare Hospital, Shenzhen, Guangdong
  - Department of Obstetrics and Gynecology, The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha, Hunan
  - Department of Obstetrics and Gynecology, Qilu Hospital of Shandong University,, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romero R, Dey SK, Fisher SJ. Preterm labor: one syndrome, many causes. Science. 2014 Aug 15;345(6198):760-5. doi: 10.1126/science.1251816. Epub 2014 Aug 14. PMID 25124429
- [Background] Boyle AK, Rinaldi SF, Norman JE, Stock SJ. Preterm birth: Inflammation, fetal injury and treatment strategies. J Reprod Immunol. 2017 Feb;119:62-66. doi: 10.1016/j.jri.2016.11.008. Epub 2016 Dec 2. PMID 28122664